CLINICAL TRIAL: NCT05898113
Title: Development of Oil with Healthy Properties Based on Corbella Olive Variety (HEVOOC)
Brief Title: Effect of the Intake of Corbella Extra Virgin Olive Oil on the Microbiota-gut-brain Axis in Healthy Adults (HEVOOC)
Acronym: HEVOOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Responsible Party: Principal Investigator, Rosa M Lamuela-Raventós, FULL PROFESSOR, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ID-20210929
Record Dates: First submitted 2023-05-17; First posted 2023-06-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Healthy Nutrition
Keywords: Extra virgin olive oil; Microbiota; Polyphenol; MGBA

STUDY DESIGN:
Intervention Model Description: 1. EXPERIMENTAL: Extra virgin olive oil (EVOO): should add 0.7 g of Corbella EVOO/ kg body weight to their usual diet per day, either raw or cooked, for one month
  2. CONTROL: Olive oil low in polyphenols (OOLP): should add 0.7 g of OOLP/ kg body weight to their usual diet per day, either raw or cooked, for one month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXTRA VIRGIN (intervention / control) (Experimental): After a 3-day run in period avoiding EVOO consumption, participants will consume a daily amount of 0.7 g EVOO / kg body weight in addition to their usual diet for 1 months. They will then have 4 weeks with their usual diet and another 3-day run in period before starting the control intervention, which consists of following their usual diet plus 0.7 g olive oil low of polyphenol (OOLP)/ kg body weight daily for one month.
  Interventions: Other: EXTRA VIRGIN OLIVE OIL; Other: OLIVE OIL LOW POLYPHENOL
- LOW POLYPHENOL (control/intervention) (Experimental): After a 3-day run-in period avoiding EVOO consumption, participants will consume a daily amount of 0.7 g of OOLP/ kg body weight in addition to their usual diet for 1 month. Then, they will have 4 weeks with their usual diet and another run in period of 3 days before starting the intervention which consists of following their usual diet plus 0.7 g of EVOO / kg body weight daily for one month.
  Interventions: Other: EXTRA VIRGIN OLIVE OIL; Other: OLIVE OIL LOW POLYPHENOL

INTERVENTIONS:
Other: EXTRA VIRGIN OLIVE OIL — Participants will consume a daily amount of extra virgin olive oil. Can consume the oil either raw or cooked
Other: OLIVE OIL LOW POLYPHENOL — Participants will consume a daily amount of olive oil low polyphenol. Can consume the oil either raw or cooked

SUMMARY:
The consumption of the improved extra virgin olive oil (EVOO) of the Corbella variety could have a beneficial effect on the microbiota-intestine-brain axis (MGBA). Olive oil contains polyphenols that are not present in other oils, notably oleocanthal and oleacein, which behave similarly to ibuprofen and have a protective effect on some neurodegenerative diseases. The polyphenols of the oil present prebiotic characteristics, at the level of the intestinal microbiota, which metabolizes them forming bioactive metabolites that can have a modulating effect on the MGBA, improving brain health. In this study, the researchers seek to identify the benefits of the consumption of Corbella variety EVOO on MGBA in healthy participants. The overall benefit of the study would be to achieve knowledge that would allow its future applicability to prevent and improve certain diseases and in general contribute to optimal health.

DETAILED DESCRIPTION:
To evaluate possible effects on MGBA, a randomized, controlled, crossover nutritional trial will be conducted. Thirty healthy adult participants (between 18 and 35 years of age, with 50% male and 50% female) will be included according to the estimated sample size. Participants will consume a daily amount of 0.7 g Corbella EVOO/kg body weight plus their normal diet (experimental intervention) and 0.7 g refined olive oil (ROO)/kg body weight plus their normal diet (control intervention) for 1 month. Biological samples (plasma, peripheral blood mononuclear cells, serum, 24-hour urine, feces and saliva) will be obtained at baseline and at the end of each trial arm.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult with Body mass index (BMI) < 30 kg/m2
* Signed informed consent

Exclusion Criteria:

* Any chronic disease (e.g. cardiovascular disease, cancer or diabetes)
* Mental disorders (e.g. depression, dementia, autism, etc.)
* Cardiovascular alterations in cholesterol,triglycerides, glucose, etc.
* Current smokers
* Repeated use of antibiotics
* Frequent use of corticoids, nonsteroidal anti-inflammatory drugs
* Repeated use of vitamins
* Volunteers with extreme eating habits (i.e. Atkins diet, very high protein diets, etc.)
* Excessive alcohol consumption (>30 g/d for males and >20 g/d for females),
* Pregnant, lactating, and postmenopausal women

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Changes in brain-derived neurotrophic factor (BDNF) after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Serum samples will be analysed for mature BDNF using a Mature BDNF Rapid ELISA kit.
Changes in the gut microbiota after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Fecal samples will be collected by the volunteers using a system for easy self-collection and stabilization of microbial DNA for gut microbiome profiling (OMNIgene - GUT). The extraction of genomic DNA from fecal samples will be carried out utilizing the DNeasy Power Kit. Subsequently, microbial profiling will employ 16 S ribosomal RNA (rRNA) sequencing to investigate microbial communities, with a specific focus on bacterial phylogeny and taxonomy.
Changes in the polyphenols and their metabolites after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Polyphenols and their metabolites derived from intestinal gut microbiota will be identified and quantified in human plasma, urine, feces, and saliva samples using high performance liquid chromatography (HPLC) - Linear Trap Quadrupole (LTQ) Orbitrap-MS/MS and HPLC-MS/MS techniques.
Changes in carotenoids and their metabolites after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Carotenoids and their metabolites derived from intestinal gut microbiota will be identified and quantified in human plasma, urine, feces, and saliva samples using high performance liquid chromatography (HPLC) - Linear Trap Quadrupole (LTQ) Orbitrap-MS/MS and HPLC-MS/MS techniques.
Changes in the short-chain fatty acids in plasma and feces samples after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  After acidifying the fecal samples with formic acid, a quantification of short-chain fatty acids will be performed using gas chromatography by direct injection according to previously described methodology (Zhao et al., 2006).
Changes in bile acids in plasma and feces samples after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Bile acids will be assayed using a validated liquid chromatography-mass spectrometry (LC-MS) method
Changes in cerebrovascular function after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Cerebrovascular function will be measured using functional magnetic resonance imaging (FMRI), a non-invasive method for assessing brain activity. FMRI maps blood oxygenation levels in the brain and estimates changes in the blood flow that depends on metabolic function and is correlated with specific brain region activities

SECONDARY OUTCOMES:
Changes in body weight after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Body weight in kilograms (kg)
Changes in body mass index (BMI) after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  BMI will be calculated as body weight (kg) divided by height (m). Weight and height will be combined to report BMI in kg/m^2
Changes in hip circumference after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  It will be measured with a tape-measure in triplicate, in centimeters (cm)
Changes in waist circumference after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  It will be measured with a tape-measure in triplicate, in centimeters (cm)
Changes in body composition after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Body fat percentage will be measured using a bioelectrical impedance analysis monitor.
Changes in blood pressure after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Diastolic and systolic blood pressure will be measured by a blood pressure monitor in triplicate.
Changes in heart rate after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Heart rate (bpm) will be measured with an automatic monitor in triplicate.
Changes in lipidic profile after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides (mg/dL) will be measured by molecular absorption spectrometry.
Changes in liver function after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP) and albumin will be assayed by immunoenzymatic methods.
Changes in glucose after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Glucose (mg/dL) will be measured by molecular absorption spectrometry.
Assessing variations in inflammatory biomarkers post-intervention for both EVOO treatments and the control group. | Baseline and after completed each intervention (1 month)
  Cytokines (pg/mL) will be assayed by immunoenzymatic methods.
Changes in inflammatory biomarkers after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Tumor necrosis factor α (TNF-α) (pg/mL) will be assayed by immunoenzymatic methods.
Changes in inflammatory biomarkers after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  C-reactive protein (CRP) (mg/dL) will be assayed by immunoenzymatic methods.
Changes in nutrients and energy intake after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  A 7-day food recall will be used. The data will be analyzed using a software called Professional Nutritional Calculation Program (PCN Pro)
Changes in quality of the diet after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Participants will fill the validated Mediterranean Diet Adherence Screener (MEDAS) questionnaire used in the PREDIMED study. This questionnaire has been validated for the Spanish population and assesses adherence to the Mediterranean diet.The MEDAS score can range from 0 to 17 and higher scores mean better outcome.
Changes in physical activity after each intervention with EVOO and the control intervention. | Baseline and after completed each intervention (1 month)
  Physical activity will be assessed with the ActiGraph® wGT3X-BT accelerometer
Changes in sleep quality after each intervention with EVOO and the control intervention | Baseline and after completed each intervention (1 month)
  Sleep quality will be assessed with the ActiGraph® wGT3X-BT accelerometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Food Sciences and Gastronomy. School of Farmacy and Food Sciences. University of Barcelona., Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No